CLINICAL TRIAL: NCT05000840
Title: Integrating Abbott Point-of-Care Technologies and the SDRI Community Scientist Model to Support HbA1c Testing Per the American Diabetes Association Guidelines for U.S. Latino Adults With or at Risk of Diabetes
Brief Title: Integrating Abbott Point-of-Care Technologies and the Community Scientist Model to Support HbA1c Testing Per ADA
Status: Active, not recruiting | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Abbott (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Kristin Castorino, DO, VP, Clinical Research and Senior Investigator, Sansum Diabetes Research Institute
Other Study IDs: CMI-IIS-002
Record Dates: First submitted 2021-07-21; First posted 2021-08-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Minority Health;; Type 2 Diabetes; Hispanic/Latino; Especialistas; Community Scientists; Community Health Workers; Social determinants of health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- HbA1c <7.5%: For participants with HbA1c ≥ 7.5%, Community Scientists will offer enrollment in existing SDRI diabetes education programs and will schedule a follow-up contact for 3 and 6 months later for repeat testing. Study participation for each participant will end upon completion of 6 month follow up.
  Interventions: Behavioral: Enrollment in existing SDRI diabetes education programs
- HbA1c ≥7.5%: For participants with HbA1c < 7.5%, Community Scientists will schedule a follow-up contact 6 months later. Study participation for each participant will end upon completion of 6 month follow up.

INTERVENTIONS:
Behavioral: Enrollment in existing SDRI diabetes education programs — Education will be based on a modification of the existing Ocho Pasos education program provided by SDRI.
  Groups: HbA1c <7.5%

SUMMARY:
In the United States, the growing Hispanic/Latino population is at high risk for type 2 diabetes and associated complications, yet underserved in healthcare and underrepresented in research. The purpose of this Sansum Diabetes Research Institute (SDRI) study is to create an HbA1c testing and support closed-loop system for U.S. Hispanic/Latino families. This loop will integrate Abbott's point-of-care (POC) technology with SDRI's Community Scientist Model to contact, test, intervene, and monitor Latinos with or at risk of type 2 diabetes for HbA1c levels. This study is built on prior work using specially trained Hispanic/Latino Community Scientists/Especialistas to support engagement with and encourage adherence to American Diabetes Association guidelines for HbA1c testing among Hispanic/Latino adults with type 2 diabetes. The study is an unblinded, nonrandomized, two arm self-controlled single center study. It is anticipated to run over 24 months and enroll 750 participants, in whom HbA1c will be measured over 6 months. This study will provide unique data on the burden of type 2 diabetes for Hispanic/Latino adults in Santa Barbara County, CA. In addition, the closed-loop approach will provide proof-of-concept evidence for scaling this approach to the larger Hispanic/Latino community to reduce the risk of poor outcomes due to type 2 diabetes and now COVID-19.

DETAILED DESCRIPTION:
Hypothesis: Adoption of the SDRI Community Scientist/Especialista model will improve adherence to ADA recommended guidelines for HbA1c testing for Hispanic/Latino adults with T2D.

Participants known to have or considered to have diabetes by the Principal Investigator (PI) will be offered enrollment in the study, and their HbA1c will be tested using the Afinion HbA1c point-of-care analyzer. The subjects will be stratified into two groups: HbA1c <7.5 and HbA1c ≥7.5%. All other potential participants (unknown diabetes diagnosis) will be tested for HbA1c as the site standard practice. All participants with HbA1c <7.5 will be followed up at 6 months; those with HbA1c ≥7.5% will be followed up at 3 months and again at 6 months post enrollment. Participants with HbA1c ≥7.5% will be invited to participate in SDRI's existing educational programs.

Therapy will be provided as per standard of care by the participant's treating physician and is out of the scope of this proposal. Those with an HbA1c at or above 7.5% will be offered diabetes education and support through the tele-health platform and/or in person. Participants not known to have diabetes but with an HbA1c result >6.4% will be referred to a local provider for further evaluation and possible diagnosis of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Hispanic/Latino individuals ≥ 18 years of age at enrollment with known or suspected T2D.
2. Ability to provide informed consent before any study-related activities. Study-related activities are any procedure that would not have been performed during normal management of the subject.
3. Based on the research staff's judgment, participant must have a good understanding, ability, and willingness to adhere to the protocol.

Exclusion Criteria:

1. Any active clinically significant physical or mental disease or disorder which, in the investigator's opinion, could interfere with the participation in the study.
2. Language barriers precluding comprehension of study activities and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be selected from Santa Barbara County and surrounding communities or satellite sites, with the help of the partnering care providers. In Santa Barbara County, Hispanic/Latino adults make up 46% of the population of almost 450,000. Data published by SDRI based on a community screening program reported that 16% of 593 Hispanic/Latino adults had an HbA1c in the diabetes range. In a cohort of Hispanic/Latino adults with known T2D, only 30% had an HbA1c less than 7%, with 31% having values greater than 9%. Currently in our Mil Familias cohort, 46% have an HbA1c above the threshold (> 7.5%) for increased risk for poor outcomes from COVID-19 (unpublished data).
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c at 3 months for participants with HbA1c ≥ 7.5% | 3 months
  HbA1c value at 3 months
HbA1c at 6 months for participants with HbA1c ≥ 7.5% | 6 months
  HbA1c value at 6 months
HcA1c at 6 months for participants with HbA1c < 7.5% | 6 months
  HbA1c value at 6 months

SECONDARY OUTCOMES:
Changes in HbA1c over time- Patient-Reported Variable #1 | 3 and/or 6 months
  Single point-in-time assessment of patient-reported variable: Socio-demographics including age, gender, race/ethnicity, insurance
Changes in HbA1c over time- Patient-Reported Variable #2 | 3 and/or 6 months
  Single point-in-time assessment of patient-reported variable: Contact Information, including smartphone ownership
Changes in HbA1c over time- Patient-Reported Variable #3 | 3 and/or 6 months
  Single point-in-time assessment of patient-reported variable: Diabetes type and duration
Changes in HbA1c over time- Patient-Reported Variable #4 | 3 and/or 6 months
  Single point-in-time assessment of patient-reported variable: Concurrent diabetes medications via visual inspection

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Thorsell, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No